CLINICAL TRIAL: NCT02270905
Title: An Open Non-comparative Clinical Investigation of a Novel Decellularised Porcine Xenograft (dCELL® Meniscus) for Partial Replacement of the Meniscus
Brief Title: Clinical Evaluation of dCELL® Meniscus for Partial Replacement of the Meniscus
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Tissue Regenix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRG-D02-01
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Knee Injuries
Keywords: meniscus; meniscectomy; decellularised; xenograft
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dCELL® Meniscus (Experimental)
  Interventions: Device: dCELL® Meniscus

INTERVENTIONS:
Device: dCELL® Meniscus — decellularised porcine xenograft

SUMMARY:
The safety and performance of dCELL® Meniscus will be evaluated in 60 patients after partial replacement of the native medial or lateral meniscus with the investigational product.

DETAILED DESCRIPTION:
The dCELL® Meniscus is a novel decellularised porcine xenograft which is processed using a patented variation of Tissue Regenix's platform dCELL® technology to render it biocompatible and free from cellular material, leaving behind an acellular biological scaffold that is safe for human implantation whilst preserving the biomechanical properties. It is indicated as a biological implant to replace parts of the native meniscus in the knee for patients who present with chronic pain following failed previous meniscus repair or partial meniscectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic pain following failed previous meniscus repair or partial meniscectomy
* Must be a stable, well aligned knee with ligament laxity of Grade II or less
* Osteoarthritis <grade 3 on the Kellgren Lawrence scale
* Patients who have given written informed consent; and are willing and able to comply with entire study procedures including rehabilitation protocol

Exclusion Criteria:

* Body Mass Index (BMI) greater than 35 kg/m2
* Treatment with any investigational drug or device within two months prior to screening
* Patients presenting with abnormal degenerative osteoarthritis of the joint
* Patients with a current ligament injury requiring immediate surgery or have had ligament surgery in the previous three months
* Patients using anticoagulants
* Patients on current immuno-suppressive or radiation therapy or having received such therapies within six months of screening
* Patients with diabetes or cardiovascular disease which precludes elective surgery
* Patients with documented renal disease or metabolic bone disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief as assessed by Visual Analog Scale (VAS) | 24 months
  Change in VAS Pain score from baseline

SECONDARY OUTCOMES:
Knee functional improvement as assessed by patient questionnaires | 24 months
  IKDC, Lysholm and KOOS score change over time

CONTACTS AND LOCATIONS:
Overall Officials: David Houlihan-Burne, Principal Investigator — The Hillingdon Hospitals NHS Foundation Trust
Locations (4):
- "Ortotrauma" Spółka Z Ograniczoną, Bialystok, Poland
- United Kingdom (3):
  - The Robert Jones & Agnes Hunt Orthopaedic Hospital NHS FOUNDATION TRUST, Oswestry, Shropshire
  - The Hillingdon Hospitals NHS FOUNDATION TRUST, Uxbridge
  - Clifton Park Hospital, York